CLINICAL TRIAL: NCT01357980
Title: A Phase IIa, Multicentre, Double Blind, Single Dose, Parallel Group, Placebo Controlled, Clinical Pilot Study to Assess the Efficacy and Safety of a Single Dose, Intra-Detrusor Injections of 750 Units of Dysport® in Subjects Suffering From Neurogenic Detrusor Overactivity Following Spinal Cord Injury or Multiple Sclerosis.
Brief Title: Neurogenic Detrusor Overactivity Following Spinal Cord Injury or Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-52-52120-155; 2010-023210-31 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Detrusor Muscle Hyperactivity
Keywords: Detrusor Muscle Overactivity
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dysport 750 U (15 injection sites) (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Placebo (15 injection sites) (Placebo Comparator)
  Interventions: Drug: Placebo
- Dysport 750 U (30 injection sites) (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Placebo (30 injection sites) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 750 U intra detrusor injection on Day 1 (single dose)
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport 750 U (15 injection sites); Dysport 750 U (30 injection sites)
Drug: Placebo — Intra detrusor injection on Day 1 (single dose)
  Arms: Placebo (15 injection sites); Placebo (30 injection sites)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a single dose of 750 U of Dysport compared to placebo for the improvement in the daily incontinence episode frequency for each administration mode in subjects suffering from neurogenic detrusor overactivity following spinal cord injury or multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject, family member or care giver was willing and able to perform clean intermittent catheterisation (CIC) for the duration of the study
* Inadequate response or refractory to anticholinergic medication
* Botulinum Toxin naive for intradetrusor injections and with no previous treatment with Botulinum Toxin of any type, within 3 months prior to study entry for any other condition
* Have a minimum of 2 incontinences per day calculated as the average daily incontinence episode frequency (IEF) over the 3 days preceding the baseline visit

Exclusion Criteria:

* Significant Baseline renal and/or urinary tract pathology
* Previous treatment with any endovesical pharmacology agent including detrusor Botulinum Toxin injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (17):
- Czechia (2):
  - Faculty Hospital Motol, Prague
  - THOMAYER Faculty Hospital, Prague
- France (11):
  - Hopital Raymond Poincaré, Garches
  - Hopital HURIET, Lille
  - Hôpital Lyon Sud -Hospices Civils de Lyon, Lyon
  - Hopital de la conception, Marseille
  - CHU Hotel Dieu, Nantes
  - Groupe Hospitalier La Pitié Salpetriere, Paris
  - Hopital Tenon, Paris
  - CMRRF Kerpape, Ploemeur
  - CHU Rouen - Hopital Charles Nicolle, Rouen
  - Nouvel Hopital civil de Strasbourg, Strasbourg
  - CHU Toulouse - Hopital Rangueil, Toulouse
- Germany (2):
  - Universitätsklinik Kiel, Kiel
  - Städtisches Klinikum Neunkirchen, Neunkirchen
- Ospedale Careggi, Florence, Italy
- NZOZ Centrum Medyczne Mazovia, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Background] Denys P, Del Popolo G, Amarenco G, Karsenty G, Le Berre P, Padrazzi B, Picaut P; Dysport Study Group. Efficacy and safety of two administration modes of an intra-detrusor injection of 750 units dysport(R) (abobotulinumtoxinA) in patients suffering from refractory neurogenic detrusor overactivity (NDO): A randomised placebo-controlled phase IIa study. Neurourol Urodyn. 2017 Feb;36(2):457-462. doi: 10.1002/nau.22954. Epub 2016 Jan 12. PMID 26756554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 22 centres in six countries (Austria, the Czech Republic, Germany, France, Italy and Poland), including 17 centres in five countries (the Czech Republic, Germany, France, Italy and Poland) which enrolled patients.
Pre-assignment Details: A screening visit was performed four to seven days prior to Baseline (Day -7 to Day -4).
  At Baseline, 47 subjects were randomised in a ratio of 5:2:5:2 to one of the four treatment groups.
Groups:
- Dysport 750 U (15 Injection Sites); Dysport 750 U (30 Injection Sites): Botulinum type A toxin (Dysport®): 750 U intra detrusor injection on day 1 (single dose)
Period: Overall Study
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Started | 16 | 7 | 17 | 7
Completed | 16 | 6 | 16 | 7
Not Completed | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Consent withdrawn | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic characteristics of the Intent to Treat (ITT) population: All randomised subjects who received at least one injection of study treatment and had an assessment for the averaged daily IEF both at Baseline and Day 84.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites) | Total
Number analyzed (Participants) | 14 | 6 | 16 | 6 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.1) | 46.5 (10.7) | 50.5 (11.1) | 40.8 (10.6) | 47.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 12 | 2 | 23
  Male | 7 | 4 | 4 | 4 | 19
Number of subjects with Spinal Cord Injury (SCI) or Multiple Sclerosis (MS) [Number; unit: participants]
  SCI | 9 | 4 | 7 | 2 | 22
  MS | 5 | 2 | 9 | 4 | 20
Number of Subjects Using Anticholinergics [Number; unit: participants] | 9 | 5 | 9 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Daily Incontinence Episode Frequency (IEF)
Time Frame: Baseline and Day 84
Population: Analysis based on number of subjects in the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: episodes per day
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
episodes per day
  Baseline | 4.21 (2.32) | 3.33 (2.87) | 3.23 (1.26) | 4.40 (1.55)
  Change from baseline to Day 84 | -3.51 (2.80) | -1.05 (2.95) | -2.86 (1.43) | -3.40 (1.49)
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the average Daily IEF change from baseline to DAY 84 using ANCOVA with the baseline average daily IEF value as covariate; Test type: Superiority or Other; p = 0.11, ANCOVA — No multiplicity adjustment applied: each test conducted at a 5% significance level; Mean Treatment Difference = -1.54, 95% CI 2-sided [-3.47 to 0.39]
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.07, ANCOVA — No multiplicity adjustment applied: each test conducted at a 5% significance level; Mean Treatment Difference = -0.61, 95% CI 2-sided [-1.27 to 0.05]

2. Secondary Outcome: Urodynamics: Maximum Cystometric Capacity
Description: Maximum Cystometric Capacity is an urodynamic parameter that indicates the volume at which a patient feels he (she) can no longer delay release of urine from the urinary bladder. Baseline urodynamics exams done at screening visit.
Time Frame: Baseline, Days 14, 42 and 84
Population: Analysis based on number (n) of subjects with a valid value in the Intent-to-Treat (ITT) population for the respective treatment groups.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
mL
  Baseline (n=14,5,16,6) | 281 (186) | 287 (112) | 288 (144) | 220 (55)
  Change from baseline to D14 (n=14,5,16,6) | 186 (160) | -36 (140) | 169 (92) | -33 (88)
  Change from baseline to D42 (n=14,6,15,6) | 163 (208) | 45 (64) | 185 (174) | 3 (94)
  Change from baseline to D84 (n=14,5,16,6) | 150 (174) | 12.5 (26) | 196 (135) | 50 (145)
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Cystometric Capacity change from baseline to DAY 14 using ANCOVA with the baseline maximum Cystometric Capacity as covariate; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = 219.5, 95% CI 2-sided [69.6 to 369.5]
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = 224.1, 95% CI 2-sided [140.9 to 307.4]
Statistical Analysis 3: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Cystometric Capacity change from baseline to DAY 42 using ANCOVA with the baseline maximum Cystometric Capacity as covariate; Test type: Superiority or Other; p = 0.09, ANCOVA; Mean Treatment Difference = 117.0, 95% CI [-20.0 to 254.0]
Statistical Analysis 4: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = 223.7, 95% CI 2-sided [94.3 to 353.1]
Statistical Analysis 5: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Cystometric Capacity change from baseline to DAY 84 using ANCOVA with the baseline maximum Cystometric Capacity as covariate; Test type: Superiority or Other; p = 0.01, ANCOVA; Mean Treatment Difference = 138.5, 95% CI 2-sided [34.7 to 242.2]
Statistical Analysis 6: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = 186.3, 95% CI 2-sided [53.2 to 319.4]

3. Secondary Outcome: Urodynamics:Maximum Detrusor Pressure
Description: Maximum Detrusor Pressure is an urodynamic parameter that is the maximum value of the pressure within the bladder which is measured during the filling phase of the urodynamic exam. Baseline urodynamics exams done at screening visit.
Time Frame: Baseline, Days 14, 42 and 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm water (cm H20)
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
cm water (cm H20)
  Baseline (n=14,5,15,6) | 59 (44) | 53 (40) | 46 (28) | 70 (23)
  Change from baseline to D14 (n=14,5,16,6) | -24 (53) | -4 (18) | -27 (22) | 27 (48)
  Change from baseline to D42 (n=14,6,15,6) | -41 (40) | -0.0 (14) | -24 (24) | 10 (42)
  Change from baseline to D84 (n=13,5,16,6) | -26 (46) | 4 (18) | -20 (23) | 12 (29)
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Detrusor Pressure change from baseline to DAY 14 using ANCOVA with the baseline Maximum Detrusor Pressure as covariate; Test type: Superiority or Other; p = 0.25, ANCOVA; Mean Treatment Difference = -23.8, 95% CI 2-sided [-66.6 to 18.9]
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = -67.1, 95% CI 2-sided [-112.9 to -21.2]
Statistical Analysis 3: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Detrusor Pressure change from baseline to DAY 42 using ANCOVA with the baseline Maximum Detrusor Pressure as covariate; Test type: Superiority or Other; p = 0.03, ANCOVA; Mean Treatment Difference = -35.1, 95% CI 2-sided [-65.6 to -4.6]
Statistical Analysis 4: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.01, ANCOVA; Mean Treatment Difference = -51.0, 95% CI 2-sided [-89.5 to -12.4]
Statistical Analysis 5: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the maximum Detrusor Pressure change from baseline to DAY 84 using ANCOVA with the baseline Maximum Detrusor Pressure as covariate; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = -32.3, 95% CI 2-sided [-53.7 to -11.0]
Statistical Analysis 6: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = -45.3, 95% CI 2-sided [-76.6 to -14.1]

4. Secondary Outcome: Physician's Global Assessment Score of Treatment Response
Description: The subject's treatment response was assessed by the physician and graded as 'markedly worse', 'much worse', 'worse', 'slightly worse', 'no change', 'slightly improved', 'improved', 'much improved', or 'markedly improved'.
Time Frame: Day 14
Population: Analysis based on number of subjects in the Intent to Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
participants
  Markedly worse | 0 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0
  Worse | 0 | 0 | 0 | 0
  Slightly worse | 1 | 1 | 0 | 1
  No change | 2 | 3 | 1 | 3
  Slightly improved | 0 | 0 | 0 | 0
  Improved | 3 | 1 | 4 | 2
  Much improved | 4 | 1 | 8 | 0
  Markedly improved | 4 | 0 | 3 | 0
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Physician's Global Assessment score at DAY 14 using a two sided Satterthwaite-Welch's t-test for independent samples; Test type: Superiority or Other; p = 0.05, Satterthwaite-Welch's t-test; Mean Treatment Difference = 1.7
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.01, Satterthwaite-Welch's t-test; Mean Treatment Difference = 2.3

5. Secondary Outcome: Physician's Global Assessment Score of Treatment Response
Description: as for outcome 4
Time Frame: Day 42
Population: Analysis based on number of subjects in the Intent to Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
participants
  Markedly worse | 0 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0
  Worse | 0 | 0 | 0 | 0
  Slightly worse | 0 | 1 | 1 | 0
  No change | 1 | 3 | 0 | 3
  Slightly improved | 0 | 0 | 0 | 0
  Improved | 3 | 1 | 4 | 3
  Much improved | 5 | 1 | 7 | 0
  Markedly improved | 5 | 0 | 4 | 0
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Physician's Global Assessment score at DAY 42 using a two sided Satterthwaite-Welch's t-test for independent samples; Test type: Superiority or Other; p = 0.01, Satterthwaite-Welch's t-test; Mean Treatment Difference = 2.3
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.01, Satterthwaite-Welch's t-test; Mean Treatment Difference = 1.8

6. Secondary Outcome: Physician's Global Assessment Score of Treatment Response
Description: as for outcome 4
Time Frame: Day 84
Population: Analysis based on number of subjects in the Intent to Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
participants
  Markedly worse | 0 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0
  Worse | 0 | 1 | 0 | 0
  Slightly worse | 0 | 0 | 0 | 0
  No change | 1 | 2 | 1 | 4
  Slightly improved | 2 | 1 | 0 | 0
  Improved | 2 | 1 | 4 | 2
  Much improved | 6 | 1 | 7 | 0
  Markedly improved | 3 | 0 | 4 | 0
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Physician's Global Assessment score at DAY 84 using a two sided Satterthwaite-Welch's t-test for independent samples; Test type: Superiority or Other; p = 0.05, Satterthwaite-Welch's t-test; Mean Treatment Difference = 1.9
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.01, Satterthwaite-Welch's t-test; Mean Treatment Difference = 2.1

7. Secondary Outcome: Quality of Life (QoL) Total Summary Score
Description: Mean Change from Baseline in Short Form (SF)-Qualiveen Questionnaire Calculated Total Score.
  The SF-Qualiveen questionnaire is a specific health related QoL questionnaire validated for urinary disorders in subjects with neurological conditions containing 8 items looking at four scales: limitations (2 items); constraints (2 items); fears (2 items) and feelings (2 items). The 8 items each having a 5-point Likert-type scale ranging from 0="Not at all" to 4="Extremely" for the first 6 items, from 0="Never" to 4="Always" for item 7 and from 0="Always" to 4="Never" for item 8. The score per scale has been calculated as the mean of the two items. In case of one missing item among the 2 items for a given scale, the score has not been calculated.
  Total score has been calculated as the mean of all the items completed among the 8 items.
  Lower scores indicate a better QoL (i.e. no limitations, fears, constraints, or negative feelings) and higher scores indicate poorer QoL.
Time Frame: Baseline, 14, 42 and 84
Population: Analysis based on number of subjects in the Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 16 | 6
score on a scale
  Baseline | 2.4 (0.7) | 2.7 (0.6) | 2.4 (0.8) | 2.3 (1.0)
  Change from baseline to D14 | -1.1 (0.9) | -0.2 (1.0) | -0.8 (0.8) | -0.5 (1.3)
  Change from baseline to D42 | -1.0 (0.8) | -0.6 (1.2) | -1.2 (0.8) | -0.6 (1.1)
  Change from baseline to D84 | -1.3 (1.0) | -0.2 (0.7) | -1.2 (0.9) | -0.7 (1.1)
Statistical Analysis 1: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Quality of Life Total Summary score change from baseline to DAY 14 using ANCOVA with the baseline Quality of Life Total Summary score as covariate; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = -1.13, 95% CI 2-sided [-1.91 to -0.35]
Statistical Analysis 2: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7, ANCOVA; Mean Treatment Difference = -0.18, 95% CI 2-sided [-1.26 to 0.90]
Statistical Analysis 3: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Quality of Life Total Summary score change from baseline to DAY 42 using ANCOVA with the baseline Quality of Life Total Summary score as covariate; Test type: Superiority or Other; p = 0.3, ANCOVA; Mean Treatment Difference = -0.52, 95% CI 2-sided [-1.56 to 0.52]
Statistical Analysis 4: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = 0.3, ANCOVA; Mean Treatment Difference = -0.48, 95% CI 2-sided [-1.47 to 0.52]
Statistical Analysis 5: Comparison: Dysport 750 U (15 Injection Sites) vs Placebo (15 Injection Sites); Comparison of the Quality of Life Total Summary score change from baseline to DAY 84 using ANCOVA with the baseline Quality of Life Total Summary score as covariate; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Treatment Difference = -1.38, 95% CI 2-sided [-2.02 to -0.73]
Statistical Analysis 6: Comparison: Dysport 750 U (30 Injection Sites) vs Placebo (30 Injection Sites); [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.4, ANCOVA; Mean Treatment Difference = -0.40, 95% CI 2-sided [-1.35 to 0.55]

8. Secondary Outcome: Pain Visual Analogue Scale (VAS) Score: Before Treatment Injection
Description: Pain assessment using the VAS. The VAS is a 100-mm (10-cm) scoring scale. Score range on VAS is from 0 to 100 where zero [0] indicates no pain and 100 indicates worst possible pain.
Time Frame: Baseline
Population: Analysis based on number of subjects in the Safety population with a valid value.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 15 | 6
mm | 2.7 (9.0) | 12.2 (21.5) | 1.3 (2.6) | 6.7 (16.3)

9. Secondary Outcome: Pain Visual Analogue Scale (VAS) Score: During Treatment Injection Procedure
Description: as for outcome 8
Time Frame: Baseline
Population: Analysis based on number of subjects in the Safety population with a valid value.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Number analyzed (Participants) | 14 | 6 | 14 | 6
mm | 13.7 (19.3) | 11.0 (19.9) | 15.8 (19.7) | 10.0 (24.5)

ADVERSE EVENTS:
Time Frame: 98 days.
Groups:
- Dysport 750 U (15 Injection Sites); Dysport 750 U (30 Injection Sites): Botulinum type A toxin (Dysport®): 750 U using different administration regimen, intra detrusor injection on day 1 (single dose)
Arm/Group | Dysport 750 U (15 Injection Sites) | Placebo (15 Injection Sites) | Dysport 750 U (30 Injection Sites) | Placebo (30 Injection Sites)
Serious Adverse Events (participants affected / at risk) | 5/16 | 0/7 | 1/17 | 0/7
Other Adverse Events (participants affected / at risk) | 7/16 | 3/7 | 11/17 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 750 U (15 Injection Sites) (N=16) | Placebo (15 Injection Sites) (N=7) | Dysport 750 U (30 Injection Sites) (N=17) | Placebo (30 Injection Sites) (N=7)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 750 U (15 Injection Sites) (N=16) | Placebo (15 Injection Sites) (N=7) | Dysport 750 U (30 Injection Sites) (N=17) | Placebo (30 Injection Sites) (N=7)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No